CLINICAL TRIAL: NCT03997071
Title: RetroBRACE - Clinical and Functional Outcomes 2 Years After Primary ACL Repair (Internal Bracing)
Acronym: RetroBRACE
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00491; ch19Jakob
Record Dates: First submitted 2019-06-12; First posted 2019-06-25 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Rupture
Keywords: ACL repair; Internal Brace Ligament Augmentation; ACL reconstruction; Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Rupture; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: functional outcome measurement — functional outcome measured in terms of joint position sense analysis, isokinetic muscle strength measurements, gait analysis, drop jump and single leg hop tests, and balance tests

SUMMARY:
The purpose of this study is to quantify 2-year postoperative clinical and functional outcomes including side-to-side differences in gait function, balance, proprioception and muscle strength in patients treated by ACL repair with Internal Brace Ligament Augmentation.

DETAILED DESCRIPTION:
Rupture of the anterior cruciate ligament (ACL) is one of the most common injuries. In recent years, arthroscopic techniques have rapidly evolved with advanced tools such as suture anchors, resolvable pins and internal bracing techniques. One of the very latest developments in internal bracing and repair for proximal ACL ruptures is the InternalBraceTM (Arthrex Inc., Naples, Florida, USA). The purpose of this study is to quantify 2-year postoperative clinical and functional outcomes including side-to-side differences in gait function, balance, proprioception and muscle strength in patients treated by ACL repair with Internal Brace Ligament Augmentation.

ELIGIBILITY:
Inclusion Criteria:

* 2 years since ACL repair and Internal Brace Ligament Augmentation

Exclusion Criteria:

* Revision surgery within 2 years after primary repair (ACL, Total or Partial Knee Arthroplasty, Joint Infection, Fracture around knee level)
* BMI > 35 kg/m2
* Previous injury and surgical procedures of the contralateral knee
* Neuromuscular disorders affecting lower limb movement
* Additional pathologies that influence the mobility of the knee joints
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated between 05/2016 and 06/2018 with ACL repair and Internal Brace Ligament Augmentation at the Clinic of Orthopaedics and Traumatology of the University Hospital Basel
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-05-07 (Actual)

PRIMARY OUTCOMES:
joint position sense Analysis (proprioception) | single time point assessment (2 years after surgery)
  Proprioception will be assessed bilaterally using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA) with an active joint position sense protocol. Participants will be positioned with hips and knees flexed at 90°. The subjects will then actively extend their knee to the target angles of 60° or 20° flexion, respectively. The subjects will be asked to remember this position. Starting from 90° flexion they will then be asked to extend their knee and reproduce the remembered target flexion angle pressing a stop button when they think they reached the angle. The difference between the perceived angle and the initial target angle will be calculated.
muscle strength | single time point assessment (2 years after surgery)
  Muscle strength will be measured bilaterally using a dynamometer (Biodex System 4 Pro: Biodex Medical Systems, Shirley, NY, USA).
gait analysis | single time point assessment (2 years after surgery)
  Instrumented gait analysis on treadmill with embedded plantar pressure plate (h/p/cosmos, Zebris FDM-T, Isny, Germany; 7168 sensors; area, 1.5 * 0.5 m; range, 1-120 N/cm2; precision, 1-120 N/cm2 ± 5%; sampling rate, 120 Hz) and on an overground walkway with two embedded force plates (Kistler force plate 9260AA6, Kistler AG, Winterthur, Switzerland; sampling rate 2400 Hz). Patients walk barefoot for 2 minutes at 0% slope at their preferred walking speed and at 1 m/s followed by walking at preferred walking speed. The treadmill speed will be increased to preferred running speed, and data for 2 minutes running will be recorded. Maximum flexion and extension angles and joint moments will be computed using the Biomove software (Stanford University).
maximum jump height (cm) | single time point assessment (2 years after surgery)
  Participants will perform three single leg hops on each leg. Maximum jump height will be determined as the highest position of the pelvis marker compared to a standing trial
Euroquol 5 Dimensions (EQ-5D-5L) | single time point assessment (2 years after surgery)
  EQ-5D-5L questionnaire measuring generic health Status; descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. As a result, a person's health status can be defined by a 5-digit number, ranging from 11111 (having no problems in all dimensions) to 55555 (having extreme problems in all dimensions).

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Muendermann, Prof. Dr. MD, Principal Investigator — Department of Orthopaedics and Traumatology Universitätsspital Basel
Locations (1):
- Department of Orthopaedics and Traumatology, University Hospital Basel, Basel, Switzerland